CLINICAL TRIAL: NCT06852261
Title: Comparison of Early Versus Late Referral for Scapular-Focused Exercise on Shoulder Function in Head and Neck Cancer Patients Following Neck Dissection
Brief Title: Early vs. Late Referral for Scapular Exercises in Shoulder Function After Neck Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202412115RINA
Record Dates: First submitted 2025-02-03; First posted 2025-02-28 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Rehabilitation
Keywords: shoulder; exercise; Head and Neck Cancer
MeSH Terms: conditions — Motor Activity; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: early (within 2 months post-surgery) and late (after 2 months post-surgery) referral groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early (within 2 months post-surgery) referral groups. (Experimental)
  Interventions: Behavioral: Scapular-focused exercise
- late (after 2 months post-surgery) referral groups (Active Comparator)
  Interventions: Behavioral: Scapular-focused exercise

INTERVENTIONS:
Behavioral: Scapular-focused exercise — Scapular-focused exercise primarily targets the trapezius muscle, 60 minutes each session, once a week for 12 weeks.
  Arms: early (within 2 months post-surgery) referral groups.
Behavioral: Scapular-focused exercise — Scapular-focused exercise primarily targets the trapezius muscle, 60 minutes each session, once a week for 12 weeks.
  Arms: late (after 2 months post-surgery) referral groups

SUMMARY:
This study aims to investigate the effects of comparing early versus late referrals for scapular-focused exercise on shoulder function in head and neck cancer patients following neck dissection.

DETAILED DESCRIPTION:
This study will recruit 30 head and neck cancer patients with spinal accessory nerve shoulder dysfunction based on the timing of referral, which will be divided into early (within 2 months post-surgery) and late (after 2 months post-surgery) referral groups. Both groups will receive conventional physical therapy (e.g., shoulder joint mobility training, electrical stimulation, or laser therapy for pain relief) and scapular-focused exercises. Scapular-focused exercise primarily targets the trapezius muscle, 60 minutes each session, once a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Age between 20 and 65 years.
2. Newly diagnosed with head and neck cancer and experiencing clinical symptoms of accessory nerve dysfunction after unilateral neck dissection, such as shoulder drooping, restricted active range of motion in shoulder abduction, or insufficient muscle strength against gravity in shoulder abduction.
3. Scapular dyskinesia, such as asymmetrical scapular movement in multiple planes.
4. Scapular asymmetry, defined as a bilateral difference of more than 1.5 cm between the inferior angle of the scapula and the spinous process of the seventh thoracic vertebra when performing 90° shoulder abduction in the scapular plane under a 1 kg load.

Exclusion Criteria：

1. Presence of distant metastasis or cancer recurrence.
2. Inability to communicate or comprehend the questionnaire.
3. History of shoulder pain within one year before neck dissection.
4. Any condition that may affect motor performance.
5. History of neuromuscular disorders or tendon pathology in the affected shoulder, other than accessory nerve dysfunction.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Active range of motion (AROM) of shoulder abduction | Baseline (before the first exercise intervention), 12 weeks of exercise intervention
  Shoulder abduction AROM is measured in degrees three times using a universal goniometer and full-circle manual protractor, with the subject supine, shoulder in lateral rotation, and palm facing anteriorly. The protractor fulcrum is placed on the anterior acromial process, one arm aligned with the midline of the sternum, and the other with the anterior midline of the humerus, while keeping the thorax immobile to prevent vertebral lateral flexion.
scapular position | Baseline (before the first exercise intervention), 12 weeks of exercise intervention
  The modified lateral scapular slide test (MLSST) measures the medio-lateral displacement of the inferior scapular angle and asymmetry at three shoulder abduction angles. The distance between the inferior scapular angle and the spinous process of the seventh thoracic vertebra is measured three times on each side using a vernier caliper, and the average difference is calculated. The MLSST is conducted in three positions: arms at the sides (position 1), hands on hips (position 2), and holding a 1 kg dumbbell at 90° shoulder abduction with maximal internal rotation in the scapular plane (position 3).

SECONDARY OUTCOMES:
ultrasonography of upper and middle trapezius morphology | Baseline (before the first exercise intervention), 12 weeks of exercise intervention
  For upper trapezius (UT) measurement, participants sit in a height-adjustable chair with back support, knees, and hips at 90°, feet on the floor, and hands resting on their thighs. The transducer is positioned parallel to the UT muscle at an oblique angle between C7 and the acromion, then moved laterally to capture the medial portion. For middle trapezius (MT) measurement, participants sit at the table edge with knees and hips at 90°, feet flat, and arms at their sides with elbows at 90° and palms down on a pillow. The transducer is placed over the middle third of a line between the acromion's posterolateral edge and the T1 spinous process, tilted forward and downward to visualize the MT's fascial borders.
electromyography signals during maximum isometric contraction of the trapezius | Baseline (before the first exercise intervention), 12 weeks of exercise intervention
  EMG signals are recorded from the upper trapezius(UT), middle trapezius (MT), and lower trapezius (LT) at standardized landmarks. MVIC is measured before testing to prevent fatigue, with participants resisting manual force in UT, MT, and LT-specific positions, each followed by a 1-minute rest. During the task, participants sit with feet flat, holding a 1 kg dumbbell at 90° shoulder abduction with maximal internal rotation. They perform three repetitions, raising the arm in 3 seconds, holding for 5 seconds, and lowering in 3 seconds, with a 60-second rest between repetitions. Normalized RMS is expressed as %MVIC by averaging EMG data from the fifth second of each repetition and normalizing it to MVIC at 90° shoulder abduction.
shoulder pain | Baseline (before the first exercise intervention), 12 weeks of exercise intervention
  Shoulder pain levels will be assessed during exercises using a 10-cm visual analog scale (VAS).
upper extremity function | Baseline (before the first exercise intervention), 12 weeks of exercise intervention
  Upper extremity function is assessed using the Taiwan version of the DASH, a reliable 30-item self-report questionnaire where higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan Univerisity Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided